CLINICAL TRIAL: NCT07290491
Title: Impact on Survival of Chaplain Provided Spiritual Care or Psychotherapy Combined With Palliative Care Versus Palliative Care Alone in Patients With Non-Curative Malignancies
Brief Title: Spiritual Care or Psychotherapy Versus Palliative Care Alone in Patients With Non-Curative Malignancies
Acronym: SPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Hanh Mai, Hematologist-Oncologist, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037917 (HMCC-BR23-001)
Record Dates: First submitted 2024-08-09; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spiritual Care or Psychotherapy/Meditation with SoC and Palliative Measures, plus Chemotherapy (Experimental): Patients will receive either individual spiritual care from a Houston Methodist Hospital chaplain or personal psychotherapy/meditation from a psychotherapist/ meditation instructor in addition to Standard of Care and Palliative Measures, plus Chemotherapy if recommended for 24 sessions (one hour per session) over 24 weeks, per patients' choice.
  Interventions: Behavioral: Chaplain-Provided Spiritual Care; Behavioral: Psychotherapy and Meditation Intervention
- Standard of Care and Palliative Measures, plus Chemotherapy (No Intervention): Patients will receive Standard of Care and palliative measures, plus chemotherapy if recommended over 24 weeks.

INTERVENTIONS:
Behavioral: Chaplain-Provided Spiritual Care — Patients will receive 24 individual, one-on-one sessions with a board -certified chaplain.
  The goal of these sessions is to elicit the spiritual, existential, and emotional issues or distress arising from your experience of cancer and draw on intrapsychic, spiritual, and narrative resources to develop a sense of meaning of your experience that is aligned with your spiritual and existential values and outlook. Rituals often function as actions to stabilize and support persons experiencing stressful or traumatic moments as well as provide structure for meaning making. The practice of rituals will be included in these sessions as a means of integrating bodily experience into reflection as well as providing a resource for ongoing spiritual support. Rituals may include prayer practices, guided imagery, use of journaling, creation of legacy items, sacred readings, poetry, or other personalized rituals.
  Arms: Spiritual Care or Psychotherapy/Meditation with SoC and Palliative Measures, plus Chemotherapy
Behavioral: Psychotherapy and Meditation Intervention — 24 individual, one-on-one psychotherapy/ meditation sessions with a licensed psychotherapist and a meditation instructor.
  Psychotherapy, or talk therapy, is an approach for addressing stresses and emotional conflicts in life by talking with a therapist. During psychotherapy, patients will be able to discuss specific challenges in your life and will work with a psychotherapist to develop helpful coping skills. Guided Visualization Meditation will be combined with psychotherapy to help you relax the body and clear the mind. Patients will be guided by an experienced instructor to cultivate a personal sense of inner calm.
  In these psychotherapy/meditation sessions you will determine the pace that you would like to follow and how deeply you wish to engage with the practice. The sessions will be interactive, and the psychotherapist/meditation instructor will respond to your needs and preferences.
  Arms: Spiritual Care or Psychotherapy/Meditation with SoC and Palliative Measures, plus Chemotherapy

SUMMARY:
This phase III clinical trial will evaluate the impact on survival of adding chaplain-provided spiritual care or psychotherapy/meditation to standard-of-care (SOC) and palliative measures, plus chemotherapy if recommended, and comparing it with SOC and palliative measures, plus chemotherapy if recommended, in patients with non-curative malignancies. The Palliative Care Department at Houston Methodist Hospital provides essential services to patients diagnosed with advanced cancer by sharing information and resources about symptom management, pain treatment and planning for the future. It is also recognized that chaplaincy-based spiritual care of patients can be a valuable part of interdisciplinary interventions in oncology.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the trial only if all of the following criteria apply

* The patient provides written informed consent for the trial.
* Male or female ≥18 years of age on the day of informed consent signing.
* Histologically confirmed metastatic disease with life expectancy of one year or less.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3.
* Willing and able to comply with the protocol for the duration of the trial including undergoing scheduled visits and interventions.

Exclusion Criteria:

Patients are excluded from the trial if any of the following criteria apply:

* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial. If a patient develops a psychiatric disorder after baseline, he/she will not be taken off the trial.
* Mobility limitations that would interfere with cooperation with the requirements of the trial.
* Confirmed positive pregnancy test in women of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2029-05-10 (Estimated); Study Completion 2030-05-10 (Estimated)

PRIMARY OUTCOMES:
To determine the overall survival (OS) of patients with non-curative malignancies | From start of intervention till the date of death, up to 30 days after completing intervention
  To determine the overall survival (OS) of patients with non-curative malignancies who receive chaplain-provided spiritual care or psychotherapy/ meditation in addition to SOC and palliative measures, plus chemotherapy if recommended.

SECONDARY OUTCOMES:
Patient-reported quality of life assessed by the FACT-G questionnaire. | Assessed at baseline and after interventions are completed, up to 24 weeks
  FACT-G (Functional Assessment of Cancer Therapy- General) Version 4. Score values range from 0 to 135. Higher score means better outcome.
Patient-reported quality of life assessed by the DASS-42 questionnaire. | Assessed at baseline and after interventions are completed, up to 24 weeks
  DASS-42 (Depression, Anxiety and Stress Scale). Score values range from 0 to 126. Higher score means worse outcome.
Patient-reported quality of life assessed by the AAQ questionnaire. | Assessed at baseline and after interventions are completed, up to 24 weeks
  AAQ (Acceptance and Action Questionnaire II). Score values range from 7 to 49. Higher score means worse outcome.
Patient-reported quality of life assessed by the ACE questionnaire. | Assessed at baseline and after interventions are completed, up to 24 weeks
  ACE (Adverse Childhood Experience). Values range from 0 if no, and 1 if yes to any question. Higher score means worse outcome.
Patient-reported quality of life assessed by the FACIT-Sp-Ex questionnaire. | Assessed at baseline and after interventions are completed, up to 24 weeks
  FACIT-Sp-Ex (Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being Expanded Version). Score values range from 0 to 92. Higher score means better outcome.
Self-reported caretaker/physician burnout as assessed by the MBI questionnaire - Section A - Burnout. | From initial assessment until final assessments are completed, every 6 months, up to 60 months
  MBI (Maslach Burnout Inventory). Section A burnout score values range from 0 to 42. Higher score means worse outcome.
Self-reported caretaker/physician burnout as assessed by the MBI questionnaire - Section B - Depersonalization. | From initial assessment until final assessments are completed, every 6 months, up to 60 months
  MBI (Maslach Burnout Inventory). Section B Depersonalization score values range from 0 to 42. Higher score means worse outcome.
Self-reported caretaker/physician burnout as assessed by the MBI questionnaire - Section C - Personal Achievement. | From initial assessment until final assessments are completed, every 6 months, up to 60 months
  MBI (Maslach Burnout Inventory). Section C Personal Achievement score values range from 0 to 48. Higher score means better outcome.
Self-reported caretaker/physician burnout as assessed by the PROMIS questionnaire. | From initial assessment until final assessments are completed, every 6 months, up to 60 months
  PROMIS (Patient-Reported Outcomes Measurement Information System -Depression and Anxiety). Depression score values range from 8 to 40. This value is t-scored and a higher score means worse outcome. Anxiety score values range from 7 to 35. This value is t-scored and a higher score means worse outcome.
Self-reported caretaker/physician burnout as assessed by the PFI questionnaire - Professional Fulfillment. | From initial assessment until final assessments are completed, every 6 months, up to 60 months
  PFI (Professional Fulfillment Index). Questions 1-6 sum values range from 0 to 24. A higher score means better outcome.
Self-reported caretaker/physician burnout as assessed by the PFI questionnaire - Burnout. | From initial assessment until final assessments are completed, every 6 months, up to 60 months
  PFI (Professional Fulfillment Index). Questions 7-16 sum values range from 0 to 40. A higher score means worse outcome.

OTHER OUTCOMES:
Measurement of circulating suppressor and effector immunocyte profiles; intracellular cytokines, enzymes and transcription factors | From pre-intervention assessments until post-intervention assessments are completed, every 4 weeks, up to 24 weeks
  Measurement of circulating suppressor and effector immunocyte profiles; intracellular cytokines, enzymes and transcription factors; systemic levels of cytokines and other soluble immune mediators, in the two arms of the trial. Correlative descriptive analysis with these and other biomarkers will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Hanh Mai, DO, Principal Investigator — Houston Methodist Neal Cancer Center
Locations (1):
- Houston Methodist Neal Cancer Center, Houston, Texas, United States